CLINICAL TRIAL: NCT05880303
Title: Effect of Nonsurgical Periodontal Therapy (NSPT) on Inflammatory Mediators, Subgingival Microbiota and Quality of Life Impacts in Rheumatoid Arthritis Subjects With Periodontitis
Brief Title: Effect of Nonsurgical Periodontal Therapy (NSPT) on Rheumatoid Arthritis Subjects With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019813-7736
Record Dates: First submitted 2023-05-03; First posted 2023-05-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis; Rheumatoid Arthritis
Keywords: periodontitis; rheumatoid arthritis; nonsurgical periodontal therapy; professional mechanical plaque removal; oral hygiene education
MeSH Terms: conditions — Periodontitis; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial with two parallel groups (intervention versus delayed treatment), with a balanced 1:1 treatment allocation and with 6 months follow-up for both groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: single-blinded parallel arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonsurgical periodontal therapy (Experimental): Subjects in the IG will be given non-surgical periodontal treatment comprising of oral hygiene instructions, scaling and root surface debridement. Scaling will be carried out with ultrasonic scaler. For root surface debridement (for sites with PPD >4mm), local anaesthetic will be administered and ultrasonic scaler and Gracey curettes will be used. The scaling and root surface debridement will be done in 2 sittings over 2 different days within a week. Oral hygiene instructions and additional supportive scaling and root surface debridement will be repeated at 3 months and 6 months if judged necessary (presence of sites with BOP and/or PPD ≥5mm).
  Interventions: Procedure: Nonsurgical periodontal therapy
- Delayed treatment (No Intervention): Oral hygiene instructions at baseline and will be repeated at 3 months and 6 months. All subjects will receive scaling and root surface debridement at the end of the 6 month trial.

INTERVENTIONS:
Procedure: Nonsurgical periodontal therapy — Oral Hygiene education, scaling and root surface debridement at baseline and 3 months
  Other Names: Professiona mechanical plaque removal and root surface instrumentation
  Arms: Nonsurgical periodontal therapy

SUMMARY:
Periodontitis (PD), a chronic inflammatory disease which results in irreversible attachment loss, bone destruction and, if left untreated, tooth loss. Rheumatoid arthritis (RA), is an autoimmune disease characterized as a chronic inflammatory disorder leading to synovial inflammation and destruction of cartilage and bone. RA and PD which are commonly seen in elderly have many similarities in terms of pathophysiology and clinical progression. Previous findings from the investigators reported that inflamed periodontal tissues of RA subjects with PD are a potential site for post translational modification of proteins as there was increase in presence of citrullinated and carbamylated proteins in gingival tissues. Autoantibodies to these proteins have been reported to be involved in loss of immune tolerance which leads to RA and its progression. Currently there are gaps in our knowledge concerning the effect of nonsurgical periodontal therapy (NSTP), comprising oral hygiene instructions, scaling and root surface debridement on presence of these autoantibodies and inflammatory outcomes of RA. It is hypothesized that reduction in periodontal inflammation may concurrently reduce the systemic inflammatory load which is responsible in perpetuating RA joint inflammation. Here, the investigators propose to perform a randomized, controlled, single-blinded study on RA subjects with stage 2 or 3 periodontitis to assess the effect of NSTP on the reduction of these autoantibodies and inflammatory mediators as well as RA related disease activity measures such as ESR, CRP and Disease Activity Score 28-joint count (DAS28). The investigators will also assess changes in subgingival microbiota associated with RA-PD in response to NSTP using next generation sequencing. This study will help determine if RA individuals could benefit from early and appropriate NSPT, thus reducing periodontal inflammation and a similar impact on RA disease could be expected. This will ultimately improve patients' quality of life and reduce societal burden related to increased patient discomfort and treatment costs.

DETAILED DESCRIPTION:
Periodontitis (PD) is a chronic inflammatory disease which results in irreversible attachment loss, bone destruction and tooth loss. The primary aetiology of PD is the dental biofilm while the host inflammatory response causes the resulting tissue damage. PD is a major oral health problem worldwide and affects about 50% of the Malaysian population with 18% having severe PD. PD has been identified by the World Health Organisation to be a significant contributor to the global burden of oral disease and is reported to be the 6th most prevalent disease globally.

Rheumatoid arthritis (RA) is an autoimmune disease characterized as a chronic inflammatory disorder leading to synovial inflammation and destruction of the cartilage and bone. The aetiology of RA is unclear, however, prior to the clinical manifestations of RA, a preclinical immunological phase shown by the identification of serum autoantibodies is seen years before the development of RA. RA has a global prevalence of 1%, is more common in females and increases with age and has a deleterious effect on joint function and quality of life.

Many studies have concluded that there is a considerable positive association between PD and RA. Our previous study has shown that the prevalence of PD in RA subjects in University of Malaya Medical Centre was 33% with 18% of the RA subjects having severe forms of PD. Both PD and RA are chronic inflammatory diseases with similar host mediated pathogenesis and commonly seen in the elderly. They share numerous characteristics and pathogenic similarities with regards to lifestyle risk factors, immuno-genetics, disease progression and tissue destruction pathways to justify the hypothesis that there is a plausible link between them.

Prior to the onset of the clinical manifestations of RA, a pre-clinical immunological phase takes place whereby autoantibodies appear in patients' sera. Currently, the most studied autoantibodies are rheumatoid factor and anti-citrullinated protein antibodies (ACPA). Citrullination, which is a common post-translational modification of arginine to citrulline, is initiated by peptidiyl arginine deiminase enzymes (PADs) that are elevated at sites of inflammation.

It has been proposed that P. gingivalis, a bacteria commonly associated with periodontitis, is capable of citrullinating proteins through the P. gingivalis peptidyl arginine deiminase (PPAD) it releases as well as being autocitrullinated. Contradictory findings have also been reported in the literature about the presence of peptidyl citrulline-specific antibodies to PPAD (anti-PPAD antibodies) in RA and PD patients.

There is also emerging evidence on the involvement of carbamylation, a different type of post-translational modification of proteins, in the pathogenesis of RA. Carbamylation is a nonenzymatic chemical reaction with cyanate that converts lysine residues to homocitrulline. Carbamylation of proteins occurs spontaneously but is increased in the presence of either urea (chronic kidney disease) or myeloperoxidase (inflammation). It leads to the formation of anti-carbamylated protein antibodies (anti-CarP). The production of anti-CarP has been associated or implicated in the pathogenesis of atherosclerosis and RA. A recent meta-analysis concluded that anti-CarP has a moderate diagnostic value in RA. Carbamylated proteins have been identified in inflamed periodontal tissues. Thus inflamed periodontal tissues may be a possible source of carbamylated protein modification that induces breakdown of immune tolerance in susceptible individuals who then progress to developing RA.

Effects of periodontal therapy in subjects with RA and PD i) Effect on the changes in periodontal inflammatory markers and RA disease activity Nonsurgical periodontal therapy (NSPT) reduces infection and periodontal inflammation through preventive measures of good oral hygiene, supra- and sub-gingival scaling and root surface debridement. Numerous studies have demonstrated the beneficial effects of NSPT towards RA disease activity and treatment outcome.

NSPT which aims to control the dental biofilm from the supra and subgingival area has been reported to aid in decreasing systemic inflammatory markers such as interleukin-1β (IL-1β), IL-6, tumour necrosis factor-α (TNF-α), matrix-metalloproteinases-8 (MMP-8), MMP-9, erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) levels in RA subjects with PD, suggesting a reduction in systemic inflammation following nonsurgical periodontal treatment. These findings were however disputed a systematic review reported that CRP and TNF-α was not significantly reduced after NSPT in RA patients. However the authors have suggested that this lack of effect in RA subjects may be due to the small sample size used in the studies or the masking of effect due to the use of disease-modifying anti-rheumatic drugs (DMARDs), leading to a low RA disease activity state.

DAS28 score is a measure of RA disease activity in RA subjects. Researchers demonstrated that non-surgical periodontal therapy led to improvements of DAS28 scores regardless of the disease activity of RA. It was also reported that there was a positive trend towards reduction of DAS28 score following NSPT.

The investigators recent findings have confirmed that inflammed periodontal tissues in RA subjects serve as a potential site of protein carbamylation and citrullination (unpublished data). Periodontal inflammation may possibly be responsible for prompting the breakdown of immune tolerance to autoantigens and progressing to RA in individuals with genetic vulnerability. It has been hypothesized the dual hit hypothesis for pathogenesis of RA being driven by citrullination or carbamylation, or both, in inflammed periodontal tissues. Significant reduction in anti-CitP levels after 1 month of NSPT has been reported. To the best of the investigators knowledge no study has looked at the effect of periodontal therapy on levels of anti-CarbP in RA subjects with PD.

In short, the evidence on the effect of NSPT in contributing to improvements of RA status is contradictory. Most of the previous studies involved only small sample sizes with short follow-up periods. Longitudinal studies with larger samples sizes are therefore needed to warrant the role of periodontal therapy in both diseases.

ii) Effect on changes in subgingival microbial diversity The most virulent bacteria associated with chronic periodontitis are Prophromonas gingivalis (P. gingivalis), Tannarella forsythia (T.forsythia), Aggregatibacter actinomycetemcomitans (A.actinomycetemcomitans) and Treponema denticola (T.denticola). Recently, new insights into the plausible aetiological link between periodonto-pathogens and RA have been reported. A mechanistic link via citrullination between P. gingivalis and its P. gingivalis peptidyl arginine deiminase (PPAD); and RA has been suggested. Using an animal model, it has been demonstrated that collagen-induced arthritis was aggravated by injecting live P. gingivalis compared to heat-killed P. gingivalis in mice. This implies that exacerbation of RA is PPAD expression dependent. Therefore, they argued that PPAD was a possible trigger of a pathogenic autoimmune response in RA.

It has been speculated that the migration of the bacterial DNA from the oral cavity to the joint could be in free DNA form. P. gingivalis DNA within the synovial fluid and synovial tissue of inflamed joints have been observed in RA subjects. Furthermore, it was also demonstrated in animal models that P. gingivalis may be able to amplify autoimmune arthritis through systemic dissemination.

Previous clinical investigations on the associations between specific oral microbiota and RA were mostly based on serological methods. Data describing the subgingival microbiota in patients with RA using next generation sequencing technology is virtually non-existent. Only one known study has looked into the oral microbiota association with RA-PD using pyro-sequencing. The investigators demonstrated that subgingival microbiota profile in patients with new-onset RA was similar to that in patients with chronic RA and healthy subjects whose PD was of comparable severity.

Clinical trials have suggested a positive influence of NSPT on the severity of RA. However, evidence regarding the effects of NSPT on the microbiological profile in RA patients is scarce since the microbiota in subgingival biofilms were not assessed in these studies. A recent study looking at the effect of NSPT on subgingival microbiological parameters have reported that counts of P. gingivalis, T. forsythia, and T. denticola decreased significantly in PD but not in the RA-PD group.

iii) Effect on changes in oral health related quality of life (OHRQoL) and health related quality of life (HRQoL) While researchers and clinicians focus on the clinical manifestations of both PD and RA, however that which is more relevant to subjects with PD, RA or both these diseases are symptoms that are not measurable with a clinician's measurement parameter. Recognition of this shortfall has yielded in the development of numerous instruments to fill this gap of knowledge. These instruments measure patient-centred quality of life (QoL) and oral health related quality of life (OHRQoL) and contribute to ideal care management providence.

One of the most widely used instrument to measure OHRQoL in patients with PD is the Oral Health Impact Profile (OHIP) which has been adapted to many different languages and validated for use in different populations with cultural diversity. The most commonly used instrument for health related quality of life (HRQoL) in RA patients is the Health Assessment Questionnaire (HAQ) which was published by the Stanford Arthritis Center in 1981. These instruments best report the disease from a patient's perspective and measures how significantly it impacts their life.

Cross-sectional studies have demonstrated that oral health has high influence on quality of life especially in subjects with PD. The investigators previous study has found that severe PD had a greater impact on OHRQoL compared to healthy subjects. The reported impacts were mainly for functional limitation and psychological discomfort dimensions. The impacts on OHRQoL was more in generalized svere PD as compared to localized disease.

The limited mobility of joints of RA patients will affect their HRQoL and may restrict them from performing adequate oral hygiene, eventually resulting in increased inflammatory activity and possibility of periodontal disease. Thus, improvement of these complications may contribute to better QOL and OHRQoL for RA patients. This has been demonstrated that at 3 months, the QOL significantly improved in diabetes subjects with periodontitis who received periodontal treatment as compared to the control group that had no treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All RA patients who fulfill the American College of Rheumatology (formerly the American Rheumatism Association) 2010 revised criteria for the classification of RA and who are unresponsive to conventional RA treatment.
2. At least 3 sites with probing pocket depths (PPD) ≥4mm and 4 sites with clinical attachment level (CAL) ≥4mm distributed in at least 2 quadrants (Papapanou et al, 2018) and will be designated as having Stage II and Stage III periodontitis
3. Patients should have a minimum of 12 teeth present.

Exclusion Criteria:

1. Patients who are on antibiotic use during the previous 3 months before study
2. Patients who have received nonsurgical periodontal treatment within 4 months before the study.
3. Patients who have any concurrent systemic or debilitating conditions such as uncontrolled diabetes.
4. Non Malaysian subjects
5. Patients who are pregnant
6. Presence of acute dental pain or infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Change in anti-carbamylated protein antibodies. | 6 months
  The anticarbamylayed protein antibody is positive when the ELISA results exceeds a cut-off value of 6ng/mL.
Differential regulation in oral bacterial proteins | 6 months
  The protein regulation will be measured using proteomic technology with PEAKS X+ software. If the proteins are detected in both test group and control group, significant results are considered if there is >2 fold change, occur in >50% of the subjects, and the p-value is <0.05. If proteins are only detected in either group, criteria to be used to consider a significant change is that the proteins are detected in >50% of the subjects in the respective group.

SECONDARY OUTCOMES:
Change in probing pocket depth (PPD) | 6 months
  Pockets less than 5 mm which do not bleed on probing
Change in Anti-citrullinated protein levels | 6 months
  Anti-citrullinated protein levels below 6.2U/ml
Change in Disease Activity Score 28-Erythrocyte sedimentation rate (DAS28-ESR) score. | 6 months
  Disease Activity Score 28-Erythrocyte sedimentation rate scores: <2.6 suggests disease remission, 2.6-3.2 suggests low disease activity, >3.2-5.1 suggests moderate disease activity, >5.1 suggest high disease activity.
Change in myeloperoxidase | 6 months
  The myeloperoxidase is positive when the ELISA results exceeds a cut-off value of 5IU/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Rathna Devi Vaithilingam, MCD(Perio), Principal Investigator — Universiti Malaya
Locations (1):
- Universiti Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of research
Access Criteria: To anyone who wishes to access the data.

REFERENCES:
- [Background] Nunez BD, Miao L, Wang Y, Nunez MM, Klein MA, Sellke FW, Ross JN, Susulic V, Paik GY, Carrozza JP, et al. Cocaine-induced microvascular spasm in Yucatan miniature swine. In vivo and in vitro evidence of spasm. Circ Res. 1994 Feb;74(2):281-90. doi: 10.1161/01.res.74.2.281. PMID 8293567
- [Background] Lee YH, Lew PH, Cheah CW, Rahman MT, Baharuddin NA, Vaithilingam RD. Potential mechanisms linking periodontitis to rheumatoid arthritis. J Int Acad Periodontol. 2019 Jul 1;21(3):99-110. PMID 31473702
- [Background] Lee YH, Baharuddin NA, Chan SW, Rahman MT, Bartold PM, Sockalingam S, Vaithilingam RD. Localisation of citrullinated and carbamylated proteins in inflamed gingival tissues from rheumatoid arthritis patients. Clin Oral Investig. 2021 Mar;25(3):1441-1450. doi: 10.1007/s00784-020-03452-9. Epub 2020 Jul 12. PMID 32656595